CLINICAL TRIAL: NCT05434312
Title: A Single-arm, Open-label, Dose Escalation and Dose Expansion Phase 1 Trial to Determine the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of TGRX-678 in Patients With Refractory or Advanced CML
Brief Title: TGRX-678 Chinese Phase I in Chronic Myelogenous Leukemia (CML) Patients
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen TargetRx, Inc. (Industry)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TGRX-678-1001
Record Dates: First submitted 2022-05-23; First posted 2022-06-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chronic Myelogenous Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TGRX-678 (Experimental): Subjects to be treated with the investigational drug TGRX-678
  Interventions: Drug: TGRX-678

INTERVENTIONS:
Drug: TGRX-678 — Participants are given TGRX-678 tablets orally at one of the dose levels as pre-determined for the dose escalation sequence.

SUMMARY:
The purpose of this single- arm, open-lable, dose escalation + dose expansion study is to evalulate the safety, tolerability, pharmacokinetic and preliminary efficacy of TGRX-678 in Chronic Myelogenous Leukemia patients who had failure with or are intolerant to TKI treatments.

DETAILED DESCRIPTION:
This is the first-in-human trial with TGRX-678 which aims to evaluate the safety profile and preliminary efficacy profile in advanced or refractory CML patients with previous failure or intolerence to TKI treatments. The primary purpose of this study is to evaluate the safety profile of TGRX-678, including determination of the maximal tolerated dose (MTD) and recommended phase II dose (RP2D), and other safety measures of the investigational drug, such as adverse events and abnormal clinical outcomes. Preliminary efficacy profile of TGRX-678 is evaluated based on the changes in peripheral blood cells and disease-associated cytogenetic markers. The safety, tolerability and efficacy profiles, along with pharmacokinetic analysis, will be assessed together to determine the optimal dose for expansion.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study with informed consent;
* 18-75 years of age at the time of screening;
* Male or female;
* Diagnosis of CML-CP by cytomorphological examination of the bone marrow, molecular biology examination, or cytogenetic testing during the screening period (according to the NCCN guidelines (NCCN, 2021);
* Received prior treatment with imatinib, dasatinib or nilotinib; patients must be intolerant or resistant to the above drugs according to MD Anderson or ELN guidelines;
* ECOG performance status ≤ 2;
* Minimum life expectancy of 3 months;
* Adequate renal function, defined as serum creatinine <1.5× upper limit of normality (ULN)
* Adequate liver function, defined as total bilirubin <1.5× ULN, AST and ALT <2.5×ULN; if liver function is compromised due to CML, AST and ALT <5×ULN;
* Adequate coagulation function, defined as PT<1.5×ULN, INR<1.5×ULN, and APTT<1.5×ULN;
* Normal pancreatic function, defined as lipase and amylase <1.5× ULN;
* Normal QTc interval, defined as ≤450 ms in males and ≤470 ms in females, as indicated by ECG screening results;
* For women with child-bearing potential, negative pregnancy test result at screening period;
* Pregnant or breast feeding and female patients of childbearing potential must agree to use effective methods of contraception.

Exclusion Criteria:

* Received TKI treatment within 7 days of first dosing of the investigational drug, or AEs related to previous treatment has not been recovered to Grade 1 or lower (except for alopecia);
* Exposure to other antineoplastic therapies and either of the following: hydroxyurea or anagrelide within 24 h prior to the first dose; interferon or immunotherapy within 14 days prior to the first dose, or any other cytotoxic chemotherapy, radiotherapy, or investigational therapy (excluding any TKI therapy) within 28 days prior to the first dose;
* Stem cell transplant < 60 days prior to the first dose, with evidence of graft versus host disease (GVHD) or GVHD requiring immunosuppressive therapy;
* Concomitant immunosuppressive therapy (other than short term corticosteroid treatment);
* Exposure to drugs related to torsade de pointes within 1 month of the screening period;
* Cytological or pathological diagnosis of active central nervous system disorder;
* CML-CP patients already achieved complete cytogenetic response;
* CML-AP patients already achieved major hematological response;
* Significant uncontrolled cardiac disease;
* Uncontrolled hypertension (Diastolic BP > 85mm Hg; Systolic > 145 mm Hg; achieved with or without medication);
* Exposure to herbal preparations or over-the-counter medications containing herbal ingredients within 2 weeks prior to the first dose;
* Severe hemorrhagic disorders unrelated to CML;
* History of grade 3-4 pancreatitis or history of alcohol abuse;
* Uncontrolled hyper-triglyceridemia (TG>450 mg/dL);
* Malabsorption syndrome or other illness that could affect oral absorption;
* Diagnosis of another primary malignancy in the past 3 years (other than non-melanoma skin cancer, cervical carcinoma in situ, or controlled prostate cancer that have been cured within 3 years;
* Invasive/extensive surgery within 14 days prior to initiating TGRX-678 therapy;
* Active clinically significant infections, including syphilis, HIV, Hepatitis B or Hepatitis C;
* Other criteria in the opinion of the investigator or the medical monitor that is unsuitable for the study, including diseases that could compromise the patients safety or the evaluation of the drugs safety or poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) | At end of Cycle 1 (each cycle is 28 days) when the posterior probability of DLT of a dose level is higher than 33%
  To determine the MTD of TGRX-678 in CML patients
Recommended phase II dose (RP2D) | At completion of the study, an average of 1.5 years
  To detemine the RP2D of TGRX-678 in CML patients for Phase II
Safety profile (DLT) | DLT: collect during Cycle 1 (28 days)
  to record and analyse subjects with dose-limiting toxicities (DLTs)
Safety profile (AEs/SAEs) | AE and SAE: through completion of the study, an average of 1.5 years
  to record and analyse subjects with adverse events (AEs) and serious adverse events (SAEs), and

SECONDARY OUTCOMES:
Hematologic Response | at screening period, weekly in Cycle 1, bi-weekly in Cycle 2 and monthly starting from Cycle 3 (each cycle is 28 days)
  To record and analyse the hematologic response of subjects. Subjects will be determined whether complete hematologic response (CHR) or no evience of leukemia (NEL) is reached.
Cytogenetic Response | at screening period, weekly in Cycle 1, bi-weekly in Cycle 2 and monthly starting from Cycle 3 (each cycle is 28 days)
  To record and analyse the cytogenetic response of subjects subjects will be determined whether partial or complete cytogenetic response (Ph+ < 35%) is reached.
Molecular Response | at screening period, weekly in Cycle 1, bi-weekly in Cycle 2 and monthly starting from Cycle 3 (each cycle is 28 days)
  To record and analyse the molecular response of subjects Subjects will be detmined whether major molecular response (BCR-ABL1 (IS) no more than 0.1%) is reached.
Plasma Cmax | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  Cmax of TGRX-678 as measured in plasma
Plasma Tmax | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  Tmax of TGRX-678 as measured in plasma
Plasma T1/2 | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  Half life of TGRX-678 as measured in plasma
Plasma AUClast | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  AUClast of TGRX-678 as measured in plasma
Plasma AUCinf | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  AUCinf of TGRX-678 as measured in plasma
Plasma Cmin | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  Cmin of TGRX-678 as measured in plasma
Plasma AUCss | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  steady state AUC of TGRX-678 as measured in plasma
Plasma Cmax,ss | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  steady state Cmax of TGRX-678 as measured in plasma
Plasma Tmax,ss | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  steady state Tmax of TGRX-678 as measured in plasma
CL | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  Clearance of TGRX-678 as measured in plasma
Vd | Day 1, 7, 21, 28 of Cycle 1, Cycle 2 Day 28 and Cycle 3 Day 28
  Volume of distribution of TGRX-678 as measured in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Qian Jiang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No